CLINICAL TRIAL: NCT05090865
Title: Dietary Potassium Liberalization With Fruit and Vegetables Versus Potassium Restriction in People With Chronic Kidney Disease (DK-Lib CKD) Trial
Brief Title: Dietary Potassium Liberalization in Pre-Dialysis Patients
Acronym: DK-LIB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Dalhousie University (Other)
Responsible Party: Principal Investigator, Dylan MacKay, Assistant Professor, University of Manitoba
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HS25191 (B2021:104)
Record Dates: First submitted 2021-10-12; First posted 2021-10-25 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Chronic Kidney Disease; Hyperkalemia
Keywords: Potassium; Nutrition
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperkalemia | interventions — Vegetables

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liberalized dietary potassium and then restricted potassium via fruit and vegetables (Other): Participants will receive weekly supplementation of higher potassium fruit and vegetables via grocery home delivery during the liberalized dietary potassium 2-week run-in and liberalized potassium treatment period, then cross-over to the restricted potassium treatment period following a 2-week washout period. Participants will receive a 30-60 minute dietary counseling session in the first week of each treatment period from a registered dietitian (RD), either in person or via videoconference, depending on regional Coronavirus disease (COVID)-19 restrictions and participant preference, which will outline the concepts of the dietary intervention. The RD will also recommend the best ways to prepare and include the fruit and vegetables into the participant's current diet.
  Interventions: Dietary Supplement: Liberalized dietary potassium via fruits and vegetables; Dietary Supplement: Standard dietary potassium restriction
- Restricted dietary potassium and then liberalized potassium via fruit and vegetables (Other): Participants will receive weekly supplementation of higher potassium fruit and vegetables via grocery home delivery during the liberalized dietary potassium 2 week run-in and then start receiving a restricted potassium treatment period, then cross-over to the liberalized potassium treatment period following a 2-week washout period. Participants will receive a 30-60 minute dietary counseling session in the first week of each treatment period from a registered dietitian (RD), either in person or via videoconference, depending on regional COVID-19 restrictions and participant preference, which will outline the concepts of the dietary intervention. The RD will also recommend the best ways to prepare and include the fruit and vegetables into the participant's current diet
  Interventions: Dietary Supplement: Liberalized dietary potassium via fruits and vegetables; Dietary Supplement: Standard dietary potassium restriction

INTERVENTIONS:
Dietary Supplement: Liberalized dietary potassium via fruits and vegetables — On the liberalized dietary potassium intervention, participants will receive groceries delivered to their houses that contain potassium rich fruit and vegetables, that contain more than 250 mg of potassium per typical serving. Participants will be instructed to incorporate the fruit and vegetables into their diet targeting a daily intake of 2000 mg of potassium a day from delivered fruit and vegetables, and a daily dietary potassium intake of 3500 mg.
Dietary Supplement: Standard dietary potassium restriction — Participants will receive weekly supplementation of lower potassium fruit and vegetables, that deliver less than 200 mg of potassium per typical serving. Participants will be instructed to incorporate the fruit and vegetables into their diet targeting a daily intake of 500 mg of K a day from the box, and a daily dietary K intake < 2000 mg. Participants will receive counselling from a registered dietician (RD) to reinforce the potassium restriction.

SUMMARY:
The study will look at the impact of the potassium content in fruits and vegetables, on serum potassium concentrations in people with Chronic Kidney Disease (CKD) using a randomized crossover design. Participants will receive home delivery of fruit and vegetables with either higher or lower potassium content in a random order. Clinical chemistry markers from blood and urine samples, blood pressure, physical functioning and health related quality of life will be assessed throughout the duration of the trial. This study will also measure their physical functioning, using a chair stand test. The results of this study could change the dietary recommendations for people with CKD related to potassium.

DETAILED DESCRIPTION:
The kidney is a primary site of potassium regulation in the body. Hyperkalemia, elevated serum potassium, occurs in approximately 10% of patients with chronic kidney disease (CKD) and is associated with elevated all-cause mortality. To minimize the risk of hyperkalemia, individuals with CKD are told to restrict dietary potassium. This recommendation is based on very-low quality evidence. Dietary potassium restrictions can negatively impact quality of life, and may put participants at risk of nutritional deficiencies so they should be based on good quality evidence. There is a need for high quality randomized controlled trials investigating the impact of dietary potassium modification on serum potassium concentrations in people with CKD.

This trial will evaluate the impact and safety of dietary potassium liberalization using fruit and vegetables on serum potassium concentrations in people with CKD. In this 16-week study, the investigators will test if changing the amount of potassium people with CKD are eating with fruits and vegetables changes the amount of potassium in their blood. The investigators will do this by providing people with fruits and vegetables that are either high or low in potassium for a period of 6 weeks. Then these same participants will be provided with fruits and vegetables that they didn't receive in the first 6 weeks, for an additional 6 weeks in what is called a randomized crossover design. In a randomized crossover design everyone gets both treatments, but the order they get them in is chosen at random, like a coin toss. Thirty participants will be recruited to this study. The investigators will measure blood potassium during the study and see if it changes due to the change in potassium in the fruit and vegetables provided. The investigators think that changing the amount of potassium that participants eat through fruit and vegetables will not lead to a different level of potassium in the participants blood, and that having higher potassium fruit and vegetables in the diet may lead to an increase in the participants quality of life. This study's results could change the dietary recommendation given to people living CKD and potentially allow them to eat a greater variety of food.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18 years or above
* Participants who have an estimated glomerular filtration rate between 15 and 45 ml/min/1.73m2
* Serum potassium concentration between 4.5 and 5.5 milliequivalent (mEq)/L
* Hemoglobin A1c ≤ 11%
* Systolic and diastolic blood pressure <160/100 mmHg
* Are registered in the multidisciplinary nephrology clinic in Winnipeg
* Able to communicate in English and provide written informed consent

Exclusion Criteria:

* Serum potassium concentration > 5.6 mEq/L, anuria, dialysis, or acute kidney injury failure in the 6 months prior to screening
* Chronic obstructive pulmonary disease that requires the participant to be on oxygen
* New York Heart Association Class 3-4 Heart symptoms or heart, liver or renal transplant
* A myocardial infarction or stroke within the last 6 months
* Unable to consume study treatments or control, such as swallowing or gastro-intestinal issues
* Currently on potassium binding therapy
* In the opinion of the investigator any medical condition, uncontrolled systemic disease or concurrent illness that would decrease the study compliance or jeopardize the safety of the participant
* Female participant who is pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in serum potassium concentrations between treatments | between endpoints of each experimental period (week 8 to week 16)
  Serum potassium at the end of the liberalize dietary potassium period compared to the end of restricted dietary potassium period

SECONDARY OUTCOMES:
Change in physical function related quality of life between treatments | between endpoints of each experimental period (week 8 to week 16)
  Participants will complete the SF-12 physical component score of the Kidney Disease Quality of Life Short Form (KDQOL-SF) questionnaire.
Change in urinary potassium between treatments | between endpoints of each experimental period (week 8 to week 16)
  total potassium concentration in mmol/L
Change in urinary sodium between treatments | between endpoints of each experimental period (week 8 to week 16)
  Total sodium concentration in mmol/L
Urinary albumin to creatinine Ratio | between endpoints of each experimental period (week 8 to week 16)
  calculated by dividing urinary albumin concentration in milligrams by urinary creatinine concentration in grams
Urinary urea | between endpoints of each experimental period (week 8 to week 16)
  Measured in mmol/L
Urinary phosphate | between endpoints of each experimental period (week 8 to week 16)
  Measured in mmol/L
Hemoglobin A1c | between endpoints of each experimental period (week 8 to week 16)
  Measure of glycosylated hemoglobin, hemoglobin A1c, expressed as a percentage
Systolic blood pressure | between endpoints of each experimental period (week 8 to week 16)
  Blood pressure will be measured in triplicate using a validated blood pressure monitor following Kidney Disease: Improving Global Outcomes (KDIGO) 2021 measurement guidelines, the average of the 2nd and 3rd measurements will be recorded.
Diastolic blood pressure | between endpoints of each experimental period (week 8 to week 16)
  Blood pressure will be measured in triplicate using a validated blood pressure monitor following KDIGO 2021 measurement guidelines, the average of the 2nd and 3rd measurements will be recorded.
Five repetition chair stand time | between endpoints of each experimental period (week 8 to week 16)
  Assessing physical functionality by asking participant to sit with arms folded in a chair and then stand up and sit down 5 times as fast as they can, time to complete is recorded.
Dietary Intake | between endpoints of each experimental period (week 8 to week 16)
  Dietary intake will be captured via triplicate dietary recall surveys using the Automated Self-Administered 24 hours Canada (ASA24, NCI, Rockville, Maryland, USA; http:// asa24. ca/)

CONTACTS AND LOCATIONS:
Overall Officials: Dylan Mackay, PhD, Principal Investigator — University of Manitoba
Locations (2):
- Canada (2):
  - Seven Oaks General Hospital Chronic Disease Innovation Centre, Winnipeg, Manitoba
  - Health Sciences Centre, Winnipeg, Manitoba

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD)may be placed in a repository if required by a journal for publication purposes. De-identified IPD may also be requested from the principle investigator.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Data will become available following the publication of the primary results manuscript.
Access Criteria: De-identified IPD may also be requested from the principle investigator upon reasonable request.

REFERENCES:
- [Derived] Iman Y, Balshaw R, Alexiuk M, Hingwala J, Cahill L, Mollard R, Tangri N, Mackay D. Dietary potassium liberalization with fruit and vegetables versus potassium restriction in people with chronic kidney disease (DK-Lib CKD): a clinical trial protocol. BMC Nephrol. 2023 Oct 13;24(1):301. doi: 10.1186/s12882-023-03354-4. PMID 37833679